CLINICAL TRIAL: NCT03659552
Title: Feasibility of Using a Percutaneous Temporary Placement of a Transvenous Phrenic Nerve Stimulator for Diaphragm Pacing Using Jugular Access
Brief Title: Percutaneous Temporary Placement of a Transvenous Phrenic Nerve Stimulator for Diaphragm Pacing Using Jugular Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN-0012
Record Dates: First submitted 2018-05-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporary diaphragmatic pacing (Experimental): There is no comparator for this study. Single site and all patients are in the treatment allocated group of temporary diaphragmatic pacing with the LIVE Catheter which is inserted via the left jugular vein.
  Interventions: Device: LIVE Catheter

INTERVENTIONS:
Device: LIVE Catheter — Placement of a temporary LIVE Catheter central venous pacing device in the left jugular vein to pace the phrenic nerves and allow recruitment of the diaphragm muscle.

SUMMARY:
Study conducted to confirm phrenic nerve stimulation using the a transvenous Phrenic Nerve Stimulator in the left jugular vein.

DETAILED DESCRIPTION:
The Lungpacer Jugular Access Feasibility System is a prototype for the Lungpacer Diaphragm Pacing Therapy System (DPTS) and consists of the LIVE Catheter, a stimulation system with a Multipole Panel Accessory, an airflow sensor and a Heart Rate Data Capture Device. The catheter is intended for inclusion in the commercial product. The stimulation system with a Multipole Panel Accessory and a Heart Rate Data Capture Device is an interim component created to enable initial safety and feasibility testing of the Lungpacer DPTS concept.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Able and willing to give informed consent or whose legally authorized representative is able and willing to give informed consent;
* Able to undergo general anesthesia (sedation, intubation, and mechanical ventilation);
* Acceptable indication for atrial septal defect closure.

Exclusion Criteria:

* Subject has an ejection fraction of < 30%
* Subject has a co-morbid illness or life expectancy < 2 years
* Subject has experienced an acute myocardial infarction within 72 hours prior to this procedure
* Subject is contraindicated for or unwilling to take aspirin or anticoagulants
* Subject is in cardiogenic shock
* Subject has other cardiovascular disease requiring open heart surgery
* Subject is known to have a demonstrated intra cardiac thrombus on echocardiography
* Subject has been treated with paralytic medications within 72 hours prior to procedure
* Subject has significant thoracic abnormalities such that placement of a left subclavian line would be difficult
* Inability to cannulate the left subclavian vein (post-consent exclusion)
* Subject has a known or suspected phrenic nerve paralysis
* Subject has co-existing temporary or implanted cardiac electrical devices such as a pacemaker or defibrillator
* Subject has an active systemic infection or local infection at or around the insertion site
* Subject is known or suspected to be pregnant or is lactating
* Subject will be unavailable for, or is unwilling to comply with, follow up requirements of the protocol
* Subject is currently enrolled in any other study of an investigational drug or device who has received treatment under that protocol with the investigational product during the 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Successful insertion of the LIVE Catheter into the left jugular vein and stimulation of phrenic nerves | through study completion, an average of 14 days
  To determine whether in an anesthetized (sedated, intubated, and mechanically ventilated) patient the LIVE Catheter can be inserted percutaneously in the left jugular vein and, via the electrical stimulator, to transvenously stimulate one or both phrenic nerves causing the diaphragm to contract

SECONDARY OUTCOMES:
Absence of device related or procedure related adverse events | through study completion, an average of 14 days
  Assess subject for adverse events status up to 48 hours post procedure

OTHER OUTCOMES:
Tidal volume assessement | during the procedure only up to 3 hours
  Generation of tidal volume upon delivery of stimulation to the phrenic nerve(s) without spontaneous or ventilator support, as measured by the ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Linda Clark, RN, Study Director — Lungpacer Medical Inc.; Adrian Ebner, MD, Principal Investigator — Italian Hospital
Locations (1):
- Italian Hospital, Asunción, Casa Zanotti, Paraguay

IPD SHARING:
Plan to Share IPD: No
Lungpacer may at any time publish the results of and information pertaining to the investigation subject only to compliance with regulatory requirements pertaining to patient protected health information

REFERENCES:
- [Background] Michalek P, Kautznerova D. Combined use of ultrasonography and neurostimulation for therapeutic phrenic nerve block. Reg Anesth Pain Med. 2002 May-Jun;27(3):306-8. No abstract available. PMID 12016605
- [Result] Escher DJ, Furman S, Solomon N, Schwedel JB. Transvenous pacing of the phrenic nerves. Am Heart J. 1966 Aug;72(2):283-4. doi: 10.1016/0002-8703(66)90456-x. No abstract available. PMID 5915563
- [Result] Escher DJ, Ashley W, Ertag W, Parker B, Furman S, Robinson G. Clinical control of respiration by transvenous phrenic pacing. Trans Am Soc Artif Intern Organs. 1968;14:192-7. No abstract available. PMID 4882945
- [Result] Eisele JH, Noble MI, Katz J, Fung DL, Hickey RF. Bilateral phrenic-nerve block in man: technical problems and respiratory effects. Anesthesiology. 1972 Jul;37(1):64-9. doi: 10.1097/00000542-197207000-00012. No abstract available. PMID 5050104
- [Result] Aubier M, Murciano D, Lecocguic Y, Viires N, Jacquens Y, Squara P, Pariente R. Effect of hypophosphatemia on diaphragmatic contractility in patients with acute respiratory failure. N Engl J Med. 1985 Aug 15;313(7):420-4. doi: 10.1056/NEJM198508153130705. PMID 3860734
- [Result] Ishii K, Kurosawa H, Koyanagi H, Nakano K, Sakakibara N, Sato I, Noshiro M, Ohsawa M. Effects of bilateral transvenous diaphragm pacing on hemodynamic function in patients after cardiac operations. Experimental and clinical study. J Thorac Cardiovasc Surg. 1990 Jul;100(1):108-14. PMID 2366549
- [Result] Allen GM, McKenzie DK, Gandevia SC, Bass S. Reduced voluntary drive to breathe in asthmatic subjects. Respir Physiol. 1993 Jul;93(1):29-40. doi: 10.1016/0034-5687(93)90065-i. PMID 8367614
- [Result] Mulvey DA, Aquilina RJ, Elliott MW, Moxham J, Green M. Diaphragmatic dysfunction in neuralgic amyotrophy: an electrophysiologic evaluation of 16 patients presenting with dyspnea. Am Rev Respir Dis. 1993 Jan;147(1):66-71. doi: 10.1164/ajrccm/147.1.66. PMID 8420434
- [Result] McKenzie DK, Allen GM, Gandevia SC. Reduced voluntary drive to the human diaphragm at low lung volumes. Respir Physiol. 1996 Aug;105(1-2):69-76. doi: 10.1016/0034-5687(96)00021-7. PMID 8897652
- [Result] Oo T, Watt JW, Soni BM, Sett PK. Delayed diaphragm recovery in 12 patients after high cervical spinal cord injury. A retrospective review of the diaphragm status of 107 patients ventilated after acute spinal cord injury. Spinal Cord. 1999 Feb;37(2):117-22. doi: 10.1038/sj.sc.3100775. PMID 10065750
- [Result] Ahn B, Beaver T, Martin T, Hess P, Brumback BA, Ahmed S, Smith BK, Leeuwenburgh C, Martin AD, Ferreira LF. Phrenic nerve stimulation increases human diaphragm fiber force after cardiothoracic surgery. Am J Respir Crit Care Med. 2014 Oct 1;190(7):837-9. doi: 10.1164/rccm.201405-0993LE. No abstract available. PMID 25271750
- [Result] Germany R, Joseph S, James K, Kao A. A novel therapeutic approach for the treatment of central sleep apnea: The remede(R) system. Cardiovasc Revasc Med. 2014 Jun;15(4):235-9. doi: 10.1016/j.carrev.2014.03.007. Epub 2014 Mar 21. PMID 24726495
- [Result] Linhart M, Nielson A, Andrie RP, Mittmann-Braun EL, Stockigt F, Kreuz J, Nickenig G, Schrickel JW, Lickfett LM. Fluoroscopy of spontaneous breathing is more sensitive than phrenic nerve stimulation for detection of right phrenic nerve injury during cryoballoon ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2014 Aug;25(8):859-865. doi: 10.1111/jce.12431. Epub 2014 May 18. PMID 24724724